CLINICAL TRIAL: NCT03156296
Title: Ultrasound Guided Transversus Abdominis Plane Block Using Dexmedetomidine and Bupivacaine in Children Undergoing Laparoscopic Orcheopexy: Randomized Controlled Trial
Brief Title: Transversus Abdominis Plane Block Using Dexmedetomidine and Bupivacaine
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, RAGAA AHMED HERDAN, Lecturer of Anesthesia and Intensive Care, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: ultrasound guided TAP block
Record Dates: First submitted 2017-05-11; First posted 2017-05-17 (Actual); Last update posted 2018-09-24 (Actual); Status verified 2018-09

CONDITIONS: Laparoscopic Orcheopexy
Keywords: transversus abdominis plane block , Dexmedetomidine
MeSH Terms: interventions — Dexmedetomidine; Bupivacaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BUPIVACAINE (Active Comparator): patients will receive ultrasound guided TAP block using 0.3 ml/kg bupivacaine (0.125%) with a maximum volume of 20 ml + 2 ml normal saline (0.9%)
  Interventions: Drug: Bupivacaine
- DEXMEDETOMIDINE (Active Comparator): patients will receive ultrasound guided TAP block using 0.3 ml/kg bupivacaine (0.125%) with a maximum volume of 20 ml + 0.25 mg/kg dexmedetomidine dissolved in 2 ml normal saline (0.9%)
  Interventions: Drug: Dexmedetomidine

INTERVENTIONS:
Drug: Dexmedetomidine — patients will receive ultrasound guided TAP block using 0.3 ml/kg bupivacaine (0.125%) with a maximum volume of 20 ml + 0.25 mg/kg dexmedetomidine dissolved in 2 ml normal saline (0.9%)
  Arms: DEXMEDETOMIDINE
Drug: Bupivacaine — patients will receive ultrasound guided TAP block using 0.3 ml/kg bupivacaine (0.125%) with a maximum volume of 20 ml + 2 ml normal saline (0.9%)
  Arms: BUPIVACAINE

SUMMARY:
Pediatric laparoscopy has been first described in 1923 by Kelling but its use has increased since last decade. A laparoscopic approach offers several advantages over an open procedures; potentially reduces the surgical stress and fluid shifts that may accompany it; in addition there is less need for postoperative analgesia, reduction of postoperative respiratory and wound complications; shortens postoperative convalescence, including an intensive care unit stay; rapid return to normal diet and decreased overall hospital stay.

Despite the minimally invasive nature, pain can be moderate to severe in the immediate postoperative period.

Inadequate control of post-operative pain leads to several unwanted adverse events ranging from patients' discomfort and prolonged immobilization to thromboembolic phenomenon and pulmonary complications.

Analgesic multimodalities were recommended to relieve the post-operative pain. Opioids although provide satisfactory analgesia, they are associated with unwanted side-effects.

Transversus abdominis plane (TAP) block is a type of peripheral nerve block that involves innervations of the anterolateral abdominal wall. It provides adequate post-operative pain relieve following various abdominal surgeries.

With the aid of ultrasound or anatomical landmark guidance, local anesthetic (LA) is injected into the transversus abdominis fascial plane, where the nerves from T6 to L1 are located.

Ultrasound TAP block is also accompanied by a good pain relief and reduced intraoperative and postoperative opioids requirements after laparoscopic surgery. In this case a bilateral TAP block is necessary because the abdominal skin incisions for the ports of laparoscopic procedure are performed on both sides.

Unfortunately, TAP block duration is limited to the effect of administered LA. Recently, adjuvant medications were added to LA to prolong the effect of TAP block. Dexmedetomidine is a selective alpha 2 (α2) adrenergic agonist with both analgesic and sedative properties. Its use with bupivacaine either epidurally or intrathecally is associated with prolongation of the LA effect.

DETAILED DESCRIPTION:
Preoperative assessment:

The day prior to surgery, all patients will undergo pre-anesthetic checkup including detailed history, thorough general, physical, systemic examination and weight of the patient. All children will be kept nil per mouth for 8 h for solids and 2 h for clear liquids.

Preparation of the patient:

* Written consent, coagulation profile, emergency resuscitation equipments including airway devices, pediatric advanced life support drugs for LA toxicity will be available.
* All patients will be premedicated with oral midazolam of 0.5 mg/kg about 20 minutes before induction of anesthesia.

Intraoperative management:

Intraoperative monitoring will include ECG, pulse oximetry, noninvasive blood pressure, capnography and temperature probe.

All patients in this study will be anesthetized by the same team of anesthesiologists and operated upon by the same surgeon who will be unaware of the study medications.

General anesthesia will be standardized for all patients in both groups using 8 MAC sevoflurane in 100% O2 with appropriate size face mask. After intravenous access securing, atropine 0.02 mg/kg and fluid bolus of 20 ml/kg will be given to offset hemodynamic effects when pneumoperitoneum is created. Endotracheal intubation with appropriate size to the patient's age will be performed after administration of 2 mg/kg propofol and 0.5 mg/kg of atracurium. After tracheal intubation, the stomach is suctioned with an orogastric tube and bladder catheterization is done in order to decrease the risk of visceral injury during trocar insertion. Controlled mechanical ventilation will be used to maintain end-tidal carbon dioxide at 35±5 mmHg. Minute ventilation will need to be increased by 20% or more to maintain normocapnia. General anesthesia will be maintained with 2-3 MAC sevoflurane delivered in 100% O2.

Patients will be placed in the supine position and TAP block will be performed under ultrasound guidance. After skin preparation, the linear ultrasound probe (high frequency probe 7-12 MHz) connected to a portable ultrasound unit( MANDRAY ) will be placed in the axial plane across the mid-axillary line midway between the costal margin and the highest point of iliac crest. A 22 G × 50 mm PAJUNK needle attached with tubing system to a syringe filled with the LA solution will be inserted in plane with the ultrasound probe and advanced until it reaches the plane between the internal oblique and transversus abdominis muscles. After careful aspiration to exclude vascular puncture, injection of the study medication will be performed leading to separation between the internal oblique and the transversus abdominis muscles which will appear as a hypoechoic space on ultrasound. This procedure will be repeated on the opposite side of the midline.

MAP, HR, SpO2 and ETCO2 will be recorded before induction of anesthesia, before block, after the block and every 10 minutes till end of surgery. Skin incision will be made 15-20 min after TAP block (Rozen et al, 2008). An increase in HR and MAP above 20% of baseline values with skin incision will be considered signs of inadequate analgesia. In these cases, fentanyl 1 μg/kg will be given intravenously, and the case will be excluded from the study.

The table position itself may need to be changed repeatedly during the operation; both the trendelenburg and the reverse trendelenburg positions are often used. Children may be placed near the foot end of the table. Accordingly, care must be taken to secure the patient to the table (e.g., using rolls of gauze and tape). Well padding of extremities should be ensured.

Restriction of the intraabdominal pressure to 6-12 mmHg in children will be recommended. These pressures have minimal effects on cardiac index. Intraoperative hypotension defined as fall in MAP by 20% from the baseline requiring a fluid bolus and bradycardia defined as a decrease in HR by 20% from the baseline value requiring atropine will be recorded. Perioperative blood loss will be replaced using crystalloids and blood as indicated.

After completion of the surgical procedure, reversal of neuromuscular blockade effect and extubation will be done after ensuring adequate orogastric suction and empting of pneumoperitonem. Bilateral air entry should be checked at the end of anesthesia. Patients will be transferred to the postanesthesia care unit (PACU).

In PACU: MAP, HR, modified CHEOPS and nausea & vomiting score will be recorded on admission to PACU, 1, 4, 8, 12, 18, 24 h postoperatively by an observer who will be unaware of the study protocol.

Postoperative pain will be measured using a modified Children's Hospital of Eastern Ontario Pain Scale (CHEOPS).

Patients with modified CHEOPS > 6 will be given rescue analgesia with 15 mg/kg paracetamol intravenously. Those with modified CHEOPS of 4-5 will be given paracetamol 15 mg/kg as suppository. Pain scores will be recorded every 10 minutes after administration of rescue analgesia to evaluate pain relief or need for further rescue analgesia. The number of children who will need postoperative rescue analgesics and the duration of analgesia that will be taken at the time when an analgesic is required will be recorded.

Patients will be discharged from the hospital when they are pain free and there is no other medical reason to admit them to a surgical ward. The parents who will be involved in the clinical trial will be invited to complete a postoperative chart with a simple pain scale (0 = no pain/child calm; 1 = minimum pain/child irritable; 2 = mild pain/child consolable; and 3 = severe pain/child inconsolable). Parents will be instructed to give their children oral ibuprofen 10 mg/kg when pain scores 2 or 3, and not more frequently than every 8 hours.

Postoperative vomiting episodes will be recorded and treated with intravenous Metoclopramide 0.5 mg/kg. Postoperative sedation will be assessed using sedation score described by Culebras et al, 2001 (1. Awake and alert. 2. Sleeping but easily arouses to voice or light touch. 3. Arouses to loud voice or shaking. 4. Arouses with painful stimuli only. 5. Unrousable).

Other postoperative complications as infection or hematoma formation will be recorded.

The parents will be asked to evaluate their satisfaction regarding pain control at the end of 24 h postoperatively through 5-point Likert scale (1 = very satisfied, 2 = satisfied, 3 = neither satisfied nor dissatisfied, 4 = dissatisfied, 5 = very dissatisfied).

ELIGIBILITY:
Inclusion Criteria:

* ASA I-II physical status patients.
* Age between 3 and 8 years.
* Children undergoing laparoscopic orcheopexy

Exclusion Criteria:

* Parent refusal
* History of developmental delay or mental retardation, which will make observational pain intensity assessment difficult
* Hypersensitivity to any local anesthetics
* Bleeding diathesis
* History of renal, hepatic, cardiac, upper or lower airway or neurological diseases
* Any sign of infection at the puncture site of the proposed block
* History of sleep apnea with which postoperative ventilation may be required

Ages: 3 Years to 8 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Enrollment: 80 (Actual)
Dates: Start 2017-06-10 (Actual); Primary Completion 2018-08-31 (Actual); Study Completion 2018-08-31 (Actual)

PRIMARY OUTCOMES:
CHEOPS | 24 hours
  postoperative pain assessment score in children

SECONDARY OUTCOMES:
Time to first analgesia | 24 hours
  Time of intravenous paracetamol requirement postoperatively
5-point Likert scale | 24 hours
  parent satisfaction score

CONTACTS AND LOCATIONS:
Locations (1):
- Assiut University Hospital, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: No